CLINICAL TRIAL: NCT02205827
Title: A Study to Determine the Inter/Intra Observer and Intra-subject Variability of Whole Blood Clotting Time Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PER977-01-005
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2014-07

CONDITIONS: Healthy
Keywords: whole blood clotting time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm (No Intervention): healthy volunteers
  Interventions: Other: Single-arm

INTERVENTIONS:
Other: Single-arm — collection of blood for assessment of whole blood clotting time
  Other Names: Whole Blood Clotting Time assessment

SUMMARY:
The purpose of the study is to characterize the distribution and sources of variability in whole blood clotting time (WBCT) measurements in human blood collected from healthy volunteers by 5 different technicians.

DETAILED DESCRIPTION:
No investigational product was administered to any subject in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated, written informed consent (Institutional Review Board [IRB]-approved informed consent form [ICF]).
2. Healthy male and female subjects aged 18 to 65 years (inclusive) with suitable veins for venipuncture. (Healthy as determined by medical history)

Exclusion Criteria:

1. Healthy subjects who do not conform to the above inclusion criteria.
2. Healthy subjects who cannot communicate reliably with the Investigator.
3. History of major bleeding or major trauma within the past 6 months
4. Healthy volunteer with a propensity to bleed (i.e. due to recent trauma, recent surgery, peptic ulcer, active or recent gastrointestinal bleeding or bleeding from hemorrhoids).
5. Significant infection or known inflammatory process within 2 weeks of screening.
6. Treatment with any investigational products or therapies within 30 days (or 5 half lives, whichever is greater) prior to screening.
7. Received non-steroidal anti-inflammatory (NSAID) or medications (including any type of anticoagulant or aspirin [ASA]) with a direct effect on hemostasis within 7 days of testing
8. Unwillingness or inability to comply with procedures required in this protocol.
9. Subjects who are concurrently enrolled in any other clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Variability in whole blood clotting time measurement | 1 day
  Assessment of variability in whole blood clotting time measurements in human blood collected from volunteers in across five technicians

CONTACTS AND LOCATIONS:
Overall Officials: James Costin, MD, Study Director — Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc.
Locations (1):
- Quintiles Phase I Services, LLC, Overland Park, Kansas, United States